CLINICAL TRIAL: NCT05625503
Title: Does Dilution of Verapamil With Normal Saline or Blood Reduce Discomfort Felt During Intraarterial Administration?
Brief Title: Dilution of Verapamil During Intraarterial Administration
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Khalil Ibrahim, Assistant Professor of Clinical Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0722
Record Dates: First submitted 2022-11-11; First posted 2022-11-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Vasospasm;Peripheral; Burning; Pain
Keywords: cardiac catheterization; intra-arterial calcium channel blockers; radial artery spasm
MeSH Terms: conditions — Paresthesia; Pain | interventions — Verapamil; Calcium Channel Blockers; Nicardipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verapamil (Active Comparator): Intra-arterial Verapamil 5 mg (2mL) diluted with 8 mL of normal saline
  Interventions: Drug: Verapamil
- Nicardipine (Placebo Comparator): Intra-arterial Nicardipine 400 mcg undiluted (8mL)
  Interventions: Drug: Nicardipine

INTERVENTIONS:
Drug: Verapamil — All patients routinely receive intra-arterial calcium channel blockers during transradial access for coronary angiography.
  Other Names: Calcium channel blocker
  Arms: Verapamil
Drug: Nicardipine — Calcium channel blocker
  Arms: Nicardipine

SUMMARY:
This study will be a randomized, single-blind, prospective trial designed to evaluate the efficacy and safety of intra-arterial (IA) Verapamil diluted with normal saline compared to undiluted IA Nicardipine during transradial access (TRA) for percutaneous coronary angiography. Patients who are 18 years or older and undergoing non-emergent percutaneous coronary angiography via TRA will be included. Patients who are non-English speaking, pregnant, or intubated will be excluded. Patients will be randomized to one of the two following groups:

1. Group 1 will receive IA Verapamil 5 mg (2mL) diluted with 8 mL of normal saline
2. Group 2 will receive IA Nicardipine 400 mcg (undiluted, 8 mL)

The investigators will document the patient's level of discomfort on the Visual Analogue Scale 30 seconds before and after administration of IA Verapamil/Nicardipine. The investigators will also document the presence of radial artery spasms.

ELIGIBILITY:
Inclusion Criteria

* English Speaking patients who are age 18 or older
* Patient must be able to provide own consent and communicate with staff
* Patient's undergoing transradial access (TRA) for the left heart catheterization (LHC)

Exclusion Criteria

* Intubated or sedated patients
* Agitated patients requiring moderate sedation prior to TRA
* Patient's undergoing femoral access for the LHC
* Non-English speaking patients
* Contraindications to Verapamil or Nicardipine: including allergies to these medications, hypotension (mean arterial pressure <65), Bradycardia (heart rate<40)
* Emergent cardiac catheterization
* Inability to obtain radial artery access
* Conversion to radial artery access from another access site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Radial Artery Spasm | approximately 30 minutes
  The investigators will document the presence or absence of radial artery spasms with either 0,1, or 2. 0 will indicate no radial artery spasms. 1 will indicate radial artery spasms that did not require a change in strategy. 2 will indicate radial artery spasms that required a change in strategy such as alternate access.
Pain Prior to Intra-arterial Calcium Channel Blocker Administration | 30 seconds prior to administration
  Pain prior to intra-arterial calcium channel blocker administration will be assessed through the Visual Analogue Pain scale (from 0 to 10).
Pain After Intra-arterial Calcium Channel Blocker Administration | 30 seconds post administration
  Pain after intra-arterial calcium channel blocker administration will be assessed through the Visual analogue Pain Scale (from 0 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Khalil Ibrahim, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided